CLINICAL TRIAL: NCT02916173
Title: Triggering of Follicular Maturation Using Human Chorionic Gonadotrophin With Gonadotrophin Releasing Hormone Agonist Versus Human Chorionic Gonadotrophin Alone in Antagonist Protocol in Assisted Reproductive Technology : a Randomized Controlled Trial
Brief Title: Triggering of Follicular Maturation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-ART
Record Dates: First submitted 2016-09-25; First posted 2016-09-27 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Increase Pregnancy Rate
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human chorionic gonadotrophin group (Experimental): Patients will receive Human chorionic gonadotrohpin injection 5000 unit
  Interventions: Drug: Recombinant Human Chorionic Gonadotrophin
- Human chorionic gonadotrophin + agonist group (Active Comparator): patients will receive both Human chorionic gonadotrophin (2500 unit) and gonadotrophin releasing hormone agonist 1mg leuprolide acetate
  Interventions: Drug: human chorionic gonadotrophin + gonadotrophin releasing hormone agonist

INTERVENTIONS:
Drug: Recombinant Human Chorionic Gonadotrophin — 250 unit intramuscular
  Other Names: Ovitrelle
  Arms: Human chorionic gonadotrophin group
Drug: human chorionic gonadotrophin + gonadotrophin releasing hormone agonist — 250 unit intramuscular + 1 mg subcutaneous
  Arms: Human chorionic gonadotrophin + agonist group

SUMMARY:
The follicular phase of the menstrual cycle involves the hourly release of gonadotropin-releasing hormone, which binds to receptors on the gonadotropes. This results in the secretion of follicle stimulating hormone and luteinizing hormone in hourly pulses that regulate follicular growth. At midcycle, rapidly rising estradiol from the dominant follicle and a small rise in progesterone lead to a gonadotrophic surge. An increase in the amplitude of Luteinizing hormone and Follicle stimulating hormone pulses initiates oocyte maturity and triggers ovulation approximately

ELIGIBILITY:
Inclusion Criteria:

1. Infertile couples wishing to do intracytoplasmic injection trial .
2. first intracytoplasmic injection trial
3. Body mass index:18-30.

5-Antral follicular count: more than 5 follicles in one ovary 6-normal, mild or moderate male factor infertility. 7- Antimullerian hormone >1 ng/ml

Exclusion Criteria:

1. Azoospermic male.
2. Body mass index more than 29.
3. Patients with endometriosis .
4. Antimullerian hormone < 1 ng/ml

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Number of M II oocytes in both groups | 24 hours

SECONDARY OUTCOMES:
Fertilization rate in each group | 3 days
Clinical pregnancy rate in each group | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No